CLINICAL TRIAL: NCT05401110
Title: IIT2021-12-Reckamp-Osi105: Phase I Study of Osimertinib With Carotuximab in Advanced, EGFR-mutated Non-Small Cell Lung Cancer
Brief Title: Study of Osimertinib With Carotuximab in Advanced, EGFR-mutated Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Karen Reckamp, MD, MS (Other)
Collaborators: Enviro Therapeutics, Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Karen Reckamp, MD, MS, Director, Division of Medical Oncology, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021-12-Reckamp-Osi105
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer
Keywords: EGFR; Osimertinib; Carotuximab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — osimertinib; carotuximab

STUDY DESIGN:
Intervention Model Description: Single arm phase I dose escalation study with expansion cohorts.
  1. Part I: Progressive disease on at least one prior EGFR TKI
  2. Part II, Cohort 1: Progressive disease on osimertinib or other prior EGFR TKIs
  3. Part II, Cohort 2: Receiving osimertinib as front line treatment for less than 12 weeks. Persistent ctDNA with EGFR mutation between weeks 6-12 from the start of osimertinib treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Osimertinib with Carotuximab (Experimental)
  Interventions: Drug: Osimertinib; Drug: Carotuximab

INTERVENTIONS:
Drug: Osimertinib — Osimertinib given by mouth daily at 40mg or 80mg depending on the starting dose level assigned per investigator. Therapy will continue until disease progression, patient withdrawal, or treatment intolerance.
  Other Names: TAGRISSO
Drug: Carotuximab — Carotuximab is administered intravenously weekly for the first 4 weeks, then every 2 weeks at 10mg/kg or 15 mg/kg depending on the starting dose level assigned per investigator. Therapy will continue until disease progression, patient withdrawal, or treatment intolerance.
  Other Names: ENV105; TRC105

SUMMARY:
The purpose of this study is to examine the combination of osimertinib and carotuximab to assess the safety and find the recommended dose for treatment of advanced EGFR-mutated non-small cell lung cancer (NSCLC). Safety and tolerability will be measured by the number of dose-limiting toxicities, according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 5, to find the maximum tolerated dose. The secondary objectives include evaluating the rate of objective response rate, duration of response, progression-free survival, and disease control rate, along with assessing biomarkers through tumor tissue and circulating tumor DNA.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV or recurrent/metastatic non-squamous NSCLC that harbors an EGFR activating mutation (Exon 21 L858R, Exon 19 deletion, Exon 18 G719X, Exon 21 L861Q, etc). Local testing for EGFR mutations is acceptable provided it was performed in a CLIA certified lab.
* Part I: Progressive disease on at least one prior EGFR TKI
* Part II, Cohort 1: Progressive disease on osimertinib or other prior EGFR TKIs
* Part II, Cohort 2: Receiving osimertinib as front line treatment for less than 12 weeks. Persistent ctDNA with EGFR mutation between weeks 6-12 from the start of osimertinib treatment.
* Age at least 18
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2
* Archival tissue from a biopsy performed after progression of disease on previous EGFR TKI or willing to consent for a fresh tumor biopsy.
* Measurable disease by RECIST 1.1.
* Patients with untreated brain metastases are allowed provided that the patient is clinically asymptomatic and stable.
* Patients must have completed prior chemotherapy ≥ 3 weeks or radiotherapy ≥ 2 weeks prior to receiving study drugs.
* If the subject's most recent line of therapy is treatment with osimertinib, then all adverse events must be resolved to Grade 2 or better
* If the subject's most recent line of therapy is any other treatment than osimertinib, then all Adverse Events must be resolved to grade 1 or better, with the exception of fatigue, alopecia and neuropathy (which must resolve to CTCAE grade 2).
* Adequate organ function
* Women of childbearing potential and men must agree to use adequate contraception while on study.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active interstitial lung disease.
* Small cell lung cancer histology.
* Other prior malignancy that might interfere with study endpoints per opinion of the investigator.
* Prior exposure to carotuximab or any CD105 targeted antibody.
* Any major surgical procedure within 2 weeks of starting therapy.
* Patients must not have a history of uncontrolled or poorly-controlled hypertension defined as SBP > 150 mmHg or DBP > 90 mmHg within 28 days prior to enrollment.
* Active bleeding or pathologic conditions that carries a high bleeding risk (e.g. gastric ulcers).
* Use of thrombolytics within 10 days prior to the first day of carotuximab.
* Known hypersensitivity to Chinese hamster ovary products or other recombinant human, chimeric, or humanized antibodies.
* A known diagnosis of Osler-Weber-Rendu syndrome.
* Ascites or pericardial or pleural effusion requiring external drainage procedures.
* New evidence of leptomeningeal disease.
* Acute cardiovascular event within the past 6 months.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
The number of adverse events and dose-limiting toxicities to find the Recommended Phase 2 Dose (RP2D) of combination of osimertinib with carotuximab in treatment of advanced, EGFR-mutated non-small cell lung cancer. | 4 weeks
  The number of adverse events are graded by NCI CTCAE v5.0. The number of these dose-limiting toxicities (DLTs) experienced within the first treatment cycle (28 days) will be assessed to determine the RP2D.

SECONDARY OUTCOMES:
Objective response rate | Assessed from baseline until the date of first documented progression, which is the end of treatment (EOT), assessed up to 2 years.
  Proportion of participants with confirmed complete response (CR) or partial response (PR) per RECIST v.1.1.
Disease control rate | Assessed from baseline until EOT, up to 2 years.
  Proportion of participants with confirmed CR, PR, or stable disease (SD) per RECIST v.1.1
Duration of response | From baseline to first documentation of PD or death, whichever came first. Assessed up to 2 years.
  Length of time from treatment response to progressive disease (PD) per RECIST v.1.1or death.
Progression free survival. | Assessed from the time of treatment initiation (C1D1) until first documentation of progression, or death due to any cause, whichever came first. Assessed up to 2 years. One treatment cycle is 28 days.
  From Cycle 1 Day 1 (C1D1) until first documentation of PD per RECIST v.1.1 or death due to any cause.
Biomarkers using tumor tissue and serial ctDNA for mutations. | From baseline until disease progression, or death, whichever came first. Assessed up to 2 years.
  ctDNA will be evaluated for genomic alterations.
Biomarkers of response to the combination using tumor tissue and serial ctDNA. | From baseline until disease progression, or death, whichever came first. Assessed up to 2 years.
  ctDNA will be evaluated to correlate with response.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Reckamp, MD, MS, Principal Investigator — Cedars-Sinai Medical Center
Locations (5):
- United States (5):
  - Cedars-Sinai Cancer at Beverly Hills (THO), Beverly Hills, California
  - Cedars-Sinai Cancer at The Angeles Clinic and Research Institute, Los Angeles, California
  - Cedars-Sinai Cancer at SOCC, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Cedars-Sinai Cancer at Hunt Cancer Center - TMPNCC, Torrance, California

IPD SHARING:
Plan to Share IPD: No